CLINICAL TRIAL: NCT04126057
Title: Myopia Assessment of Two Manufacturing Processes for Myopia Management Lenses (MAPLE)
Brief Title: Myopia Assessment of Two Manufacturing Processes
Acronym: MAPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRO-1908-001
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Juvenile Myopia
Keywords: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DOT Spectacle Lenses using Manufacturing Method A (Experimental): Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method A
  Interventions: Device: SightGlass Vision DOT Spectacle Lenses
- DOT Spectacle Lenses using Manufacturing Method B (Experimental): Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method B
  Interventions: Device: SightGlass Vision DOT Spectacle Lenses

INTERVENTIONS:
Device: SightGlass Vision DOT Spectacle Lenses — Subjects randomized to test vs control, left eyes and right eyes
  Other Names: SightGlass Vision

SUMMARY:
Randomized, controlled, multisite, subject- and observer-masked, contralateral clinical trial of 6-month duration to compare two SightGlass Vision Diffusion Optics Technology (DOT) spectacle lens manufacturing processes in reducing the progression of juvenile myopia.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 and 14 years old (inclusive) with myopia
* Best corrected visual acuity by manifest refraction of +0.10 logMAR (20/25 Snellen equivalent) or better in each eye
* Difference in spherical equivalent power between the two eyes (anisometropia based on manifest refraction) must be less than or equal to 0.75 D

Exclusion Criteria:

* Current use of any myopia control treatment such as atropine, multifocal contact lenses, or orthokeratology (NOTE: Prior bilateral usage acceptable as long as treatment stopped at least 6 months before screening visit. Any subject with a history of unilateral myopia control treatment is excluded.)
* Any ocular or systemic conditions that could influence refractive development or status [e.g., keratoconus, congenital glaucoma, ocular trauma, diabetes, Marfan syndrome or other connective tissue disorder, Down's syndrome, family history of poor night vision (to prevent against enrolling subjects with congenital stationary night blindness)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rappon, OD, MS, FAAO, Study Chair — SightGlass Vision, Inc.
Locations (5):
- United States (5):
  - Sabal Eye Care, Longwood, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Advanced Eyecare PC, Raytown, Missouri
  - SUNY School of Optometry, New York, New York
  - William J Bogus, OD, FAAO, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- DOT Spectacle Lenses Test: Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method A
  SightGlass Vision DOT Spectacle Lenses: Subjects randomized to test vs control, left eyes and right eyes
- DOT Spectacle Lenses Control: Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method B
  SightGlass Vision DOT Spectacle Lenses: Subjects randomized to test vs control, left eyes and right eyes
Period: Overall Study
Arm/Group | DOT Spectacle Lenses Test | DOT Spectacle Lenses Control
Started | 50; 50 Eyes | 50; 50 Eyes
Completed | 47; 47 Eyes | 46; 46 Eyes
Not Completed | 3; 3 Eyes | 4; 4 Eyes

BASELINE CHARACTERISTICS:
Population: This was a contralateral eye study of 50 participants in which both eyes were enrolled. In the analysis set, each group has 43 eyes with a total of 43 participants.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | DOT Spectacle Lenses Test | DOT Spectacle Lenses Control | Total
Number analyzed (Participants) | 43 | 43 | 43
Number analyzed (Eyes) | 43 | 43 | 86
Age, Categorical [Count of Units; unit: Eyes]
  <=18 years | 43 | 43 | 86
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.67 (2.073) | 11.67 (2.073) | 11.67 (2.073)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 21 | 21 | 42
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Units; unit: Eyes]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 5 | 5 | 10
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 43 | 43 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change in Axial Length Progression From Baseline
Description: Change in axial length progression over time between DOT spectacle lenses manufactured by method A versus method B Axial length progression is defined as an axial length elongation that is attributable to myopia.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Groups:
- DOT Spectacle Lenses Using Test: Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method A
  SightGlass Vision DOT Spectacle Lenses: Subjects randomized to test vs control, left eyes and right eyes
- DOT Spectacle Lenses Using Control: Single vision, impact-resistant spectacles using SightGlass Vision DOT spectacle lenses, manufacturing method B
  SightGlass Vision DOT Spectacle Lenses: Subjects randomized to test vs control, left eyes and right eyes
Arm/Group | DOT Spectacle Lenses Using Test | DOT Spectacle Lenses Using Control
Number analyzed (Participants) | 43 | 43
Number analyzed (Eyes) | 43 | 43
mm | 0.046 (0.139) | 0.047 (0.128)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DOT Spectacle Lenses Using Test | DOT Spectacle Lenses Using Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04126057/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04126057/SAP_001.pdf